CLINICAL TRIAL: NCT06484426
Title: The Goal Attainment Scaling in Down Syndrome-associated Alzheimer's Disease (DS-AD) Sub-study
Brief Title: Goal Attainment Scaling (GAS) Sub-Study
Status: Completed | Type: Observational
Sponsor: LuMind IDSC Foundation (Other)
Collaborators: Ardea Outcomes Inc. (Unknown); Pentara (Unknown)
Responsible Party: Sponsor
Other Study IDs: LIFE-DSR-GAS DS-AD
Record Dates: First submitted 2024-03-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer's Disease in Down Syndrome
Keywords: Down Syndrome; Alzheimer's Disease
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an optional sub-study that will enroll participants from LIFE-DSR parent protocol. The aim is to assess change over 16 months in individuals with Down syndrome through individualized goals set by their caregivers. This sub-study also aims to assess the feasibility of Goal Attainment Scaling in the DS-AD population.

DETAILED DESCRIPTION:
People with Down syndrome are living longer. A longer life increases the chances of age-related risks of developing Alzheimer's disease and other forms of dementia. There is also growing evidence that people with Down syndrome respond differently to treatment than people without Down syndrome. This creates an important need to create a way to identify and follow changes in thinking and behavior as people with Down syndrome age and start to experience symptoms of dementia. Here, the investigators are testing a new method to monitor changes (in thinking and behavior) called goal attainment scaling.

During this study, the participant will be asked to take part in a goal attainment scaling interview, which means working with a clinical rater (the participant's health care provider or other study team) to identify personally meaningful goals to follow for the study. "Goals" are based on symptoms or challenges experienced by the person for whom cares for the participant with Down Syndrome. The identified goals may be related to potential early signs and symptoms of Alzheimer's disease. These goals will then be reviewed at 2 time-points over the next 16 months. The investigators want to learn whether this type of interview can help the investigators understand what symptoms or challenges are important to the participant and whether this type of interview can help the investigators understand how these might change over time. The investigators also want to hear the participant's feedback about the participant's experience with goal attainment scaling at the end of the sub-study.

The investigators will be asking about 45 participants to take part in this study.

This study is observational and does not test a study drug.

ELIGIBILITY:
Inclusion Criteria:

The participant with DS and caregiver must be currently enrolled in the LIFE-DSR parent protocol.

The participant with DS must be age 35 years or older.

Both the participant with DS, or LAR, and their caregiver must be able to understand and be willing to sign written informed consent.

In the opinion of the Investigator, a participant's caregiver must have frequent interaction with the participant on a regular basis, agree to participate in clinic and remote visits, be able to provide accurate responses to questions about the participant with DS, and be capable of facilitating participation in the study visits.

Participant with DS and caregiver must be capable of reliably completing all study assessments at each time-point.

The caregiver must be able to converse in English.

Exclusion Criteria:

Unable to complete trial procedures or adhere to the schedule of study assessments, in the opinion of the site PI.

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Males and females, aged 35 and older, with a diagnosis of DS. Must be enrolled in the LIFE-DSR (the parent study to the GAS sub-study)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | 16 months
  Patient centered outcome measure aiming to assess change in individuals with Down syndrome through individualized goals set by their caregivers. This sub-study also aims to assess the feasibility of Goal Attainment Scaling in the DS-AD population.
  GoalNav® DS-AD Instrument
  This is a web-based platform developed by Ardea Outcomes with a DS-AD menu of 58 symptoms/challenges developed in collaboration with LuMind IDSC Foundation. This instrument is intended to track pre-dementia and dementia symptoms over time, including behaviors and other challenges common in adults with DS-AD.
  The goal scale is a 5-point scale. Minimum value is 1 maximum value is 5
  No indicators of what higher or lower scores mean.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, San Diego, San Diego, California
  - Advocate Health, Park Ridge, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Case Western Reserve University School of Medicine, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No